CLINICAL TRIAL: NCT02536989
Title: Comparison of High Dose Infusion and Low Dose Bolus Intravenous Omeprazole for Treatment of Bleeding Ulcer With Adherent Clot
Brief Title: Different Dose of Intravenous Omeprazole to Treat Bleeding Ulcer With Adherent Clot
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tzong-Hsi Lee, M.D., Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FEMH-96-C009
Record Dates: First submitted 2009-02-06; First posted 2015-09-01 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2010-08

CONDITIONS: Peptic Ulcer; Hemorrhage
Keywords: peptic ulcer bleeding; blood clot; dose
MeSH Terms: conditions — Peptic Ulcer; Hemorrhage; Peptic Ulcer Hemorrhage; Thrombosis | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): receive high dose PPI treament with intravenous omeprazole 80 mg stat and then 8mg/hr infusion for 3 days
  Interventions: Drug: omeprazole
- 2 (Active Comparator): receive usual dose PPI treatment with ntravenous omeprazole 40 mg stat and then 40 mg q12h for 3 days
  Interventions: Drug: omeprazole

INTERVENTIONS:
Drug: omeprazole — receive intravenous omeprazole 80 mg stat and then 8mg/hr infusion for 3 days
  Other Names: Losec, iv, high dose
  Arms: 1
Drug: omeprazole — receive intravenous omeprazole 40 mg stat and then 40 mg q12h for 3 days
  Other Names: Losec, iv, usual dose
  Arms: 2

SUMMARY:
The investigators will include those patients with adherent clot on gastric or duodenal ulcers after endoscopic confirmation After receiving well explanation and giving written consent, they are enrolled and will be allocated to 2 groups randomly. Those in the first group will receive intravenous omeprazole 40 mg stat and then 40 mg q12h. Those in the second group will receive intravenous omeprazole 80 mg stat and then 8mg/hr infusion. The patients in both groups will receive intravenous omeprazole for 3 days and then oral esomeprazole qd for further treatment of peptic ulcer.

The investigators define rebleeding during admission and within 30 days as primary end points and define surgical intervention for ulcer bleeding, transfusion amount and hospitalization days after allocation as secondary end points.

DETAILED DESCRIPTION:
The investigators will include those patients with adherent clot on gastric or duodenal ulcers after endoscopic confirmation and exclusion of other possible bleeder. Adherent clot is defined that still stays on the ulcer after 200 ml normal saline irrigation (4 times of irrigation with 50 ml syringe). After receiving well explanation and giving written consent, they are enrolled and will be allocated to 2 groups randomly. Those in the first group will receive intravenous omeprazole 40 mg stat and then 40 mg q12h. Those in the second group will receive intravenous omeprazole 80 mg stat and then 8mg/hr infusion. The patients in both groups will receive intravenous omeprazole for 3 days and then oral esomeprazole qd for further treatment of peptic ulcer. The investigators will record the basic data of these patients including age, sex, use of NSAID or anit-coagulant, concomitant major diseases; clinical data including Hb, Plt, PT, the lowest systolic pressure before allocation and heart rate at the same time, shock status, transfusion amount before allocation; endoscopic findings including the location & size of ulcer, size of clot, existence of fresh blood in stomach or duodenum. The investigators will monitor the events of rebleeding during admission and within 30 days, surgery for ulcer bleeding and mortality within 30 days and record the amount of transfusion and hospitalization days after allocation. When rebleeding is suspected , those patient will receive endoscopic examination and appropriate therapy. Further treatment with surgical or angiographic intervention is decided by the attending physicians.These patients will be monitored during admission (2 weeks in average)and then followed up in GI outpatient clinics.

The investigators define rebleeding during admission and within 30 days as primary end points. Rebleeding is defined as the one of the clinical manifestations occurring 6 hours after allocation: 1.hematemesis or bloody stool 2. tarry stool and hemodynamic change (systolic pressure less than 90 mmHg, or heart more than 110 beats per minute ) 3. decrease of Hb more than 2g/dl within 24 hours after elevation of Hb to 10 g/dl with transfusion. The investigators define surgical intervention for ulcer bleeding, transfusion amount and hospitalization days after allocation as secondary end points.

ELIGIBILITY:
Inclusion Criteria:

* We will include those patients with adherent clot, more than 5 mm, on gastric or duodenal ulcers after endoscopic confirmation and exclusion of other possible bleeder. Adherent clot is defined that still stays on the ulcer after 200 ml normal saline irrigation (4 times of irrigation with 50 ml syringe).

Exclusion Criteria:

* ulcer with active bleeding, suspected malignant ulcer, patients with age less than 18 years old, or allergy to omeprazole

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
rebleeding rate within 30 days after allocation | within 30 days after allocation

SECONDARY OUTCOMES:
blood transfusion units needed within 30 days after allocation | within 30 days after allocation

CONTACTS AND LOCATIONS:
Overall Officials: Tzong-Hsi Lee, M.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Martins NB, Wassef W. Upper gastrointestinal bleeding. Curr Opin Gastroenterol. 2006 Nov;22(6):612-9. doi: 10.1097/01.mog.0000245542.95408.5d. PMID 17053438
- [Background] Rollhauser C, Fleischer DE. Nonvariceal upper gastrointestinal bleeding. Endoscopy. 2004 Jan;36(1):52-8. doi: 10.1055/s-2004-814114. PMID 14722856
- [Background] Jung HK, Son HY, Jung SA, Yi SY, Yoo K, Kim DY, Moon IH, Lee HC. Comparison of oral omeprazole and endoscopic ethanol injection therapy for prevention of recurrent bleeding from peptic ulcers with nonbleeding visible vessels or fresh adherent clots. Am J Gastroenterol. 2002 Jul;97(7):1736-40. doi: 10.1111/j.1572-0241.2002.05780.x. PMID 12135028
- [Background] Bleau BL, Gostout CJ, Sherman KE, Shaw MJ, Harford WV, Keate RF, Bracy WP, Fleischer DE. Recurrent bleeding from peptic ulcer associated with adherent clot: a randomized study comparing endoscopic treatment with medical therapy. Gastrointest Endosc. 2002 Jul;56(1):1-6. doi: 10.1067/mge.2002.125365. PMID 12085028
- [Background] Sung JJ, Chan FK, Lau JY, Yung MY, Leung WK, Wu JC, Ng EK, Chung SC. The effect of endoscopic therapy in patients receiving omeprazole for bleeding ulcers with nonbleeding visible vessels or adherent clots: a randomized comparison. Ann Intern Med. 2003 Aug 19;139(4):237-43. doi: 10.7326/0003-4819-139-4-200308190-00005. PMID 12965978
- [Background] Sheu BS, Chi CH, Huang CC, Kao AW, Wang YL, Yang HB. Impact of intravenous omeprazole on Helicobacter pylori eradication by triple therapy in patients with peptic ulcer bleeding. Aliment Pharmacol Ther. 2002 Jan;16(1):137-43. doi: 10.1046/j.1365-2036.2002.01137.x. PMID 11856088
- [Background] Lin HJ, Lo WC, Cheng YC, Perng CL. Role of intravenous omeprazole in patients with high-risk peptic ulcer bleeding after successful endoscopic epinephrine injection: a prospective randomized comparative trial. Am J Gastroenterol. 2006 Mar;101(3):500-5. doi: 10.1111/j.1572-0241.2006.00399.x. PMID 16542286
- [Background] Lau JY, Leung WK, Wu JC, Chan FK, Wong VW, Chiu PW, Lee VW, Lee KK, Cheung FK, Siu P, Ng EK, Sung JJ. Omeprazole before endoscopy in patients with gastrointestinal bleeding. N Engl J Med. 2007 Apr 19;356(16):1631-40. doi: 10.1056/NEJMoa065703. PMID 17442905
- [Background] Swain CP, Kirkham JS, Salmon PR, Bown SG, Northfield TC. Controlled trial of Nd-YAG laser photocoagulation in bleeding peptic ulcers. Lancet. 1986 May 17;1(8490):1113-7. doi: 10.1016/s0140-6736(86)91835-0. PMID 2871378
- [Background] Kahi CJ, Jensen DM, Sung JJ, Bleau BL, Jung HK, Eckert G, Imperiale TF. Endoscopic therapy versus medical therapy for bleeding peptic ulcer with adherent clot: a meta-analysis. Gastroenterology. 2005 Sep;129(3):855-62. doi: 10.1053/j.gastro.2005.06.070. PMID 16143125
- [Background] Jensen DM, Kovacs TO, Jutabha R, Machicado GA, Gralnek IM, Savides TJ, Smith J, Jensen ME, Alofaituli G, Gornbein J. Randomized trial of medical or endoscopic therapy to prevent recurrent ulcer hemorrhage in patients with adherent clots. Gastroenterology. 2002 Aug;123(2):407-13. doi: 10.1053/gast.2002.34782. PMID 12145792
- [Background] Laine L, Freeman M, Cohen H. Lack of uniformity in evaluation of endoscopic prognostic features of bleeding ulcers. Gastrointest Endosc. 1994 Jul-Aug;40(4):411-7. doi: 10.1016/s0016-5107(94)70202-0. PMID 7926529
- [Background] Lau JY, Sung JJ, Chan AC, Lai GW, Lau JT, Ng EK, Chung SC, Li AK. Stigmata of hemorrhage in bleeding peptic ulcers: an interobserver agreement study among international experts. Gastrointest Endosc. 1997 Jul;46(1):33-6. doi: 10.1016/s0016-5107(97)70206-2. PMID 9260702
- [Background] Swain CP, Storey DW, Bown SG, Heath J, Mills TN, Salmon PR, Northfield TC, Kirkham JS, O'Sullivan JP. Nature of the bleeding vessel in recurrently bleeding gastric ulcers. Gastroenterology. 1986 Mar;90(3):595-608. doi: 10.1016/0016-5085(86)91113-3. PMID 3943691
- [Background] Laine L, Peterson WL. Bleeding peptic ulcer. N Engl J Med. 1994 Sep 15;331(11):717-27. doi: 10.1056/NEJM199409153311107. No abstract available. PMID 8058080
- [Background] Katschinski B, Logan R, Davies J, Faulkner G, Pearson J, Langman M. Prognostic factors in upper gastrointestinal bleeding. Dig Dis Sci. 1994 Apr;39(4):706-12. doi: 10.1007/BF02087411. PMID 7908623
- [Background] Consensus conference: Therapeutic endoscopy and bleeding ulcers. JAMA. 1989 Sep 8;262(10):1369-72. No abstract available. PMID 2668576